CLINICAL TRIAL: NCT02259777
Title: Influence of Food on the Bioavailability of 80 mg Telmisartan/10 mg Amlodipine Fixed Dose Combination in Healthy Male and Female Volunteers. An Open-label, Randomised, Single-dose, Two Period, Crossover Study
Brief Title: Bioavailability of Telmisartan/Amlodipine Fixed Dose Combination in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1235.12
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — telmisartan amlodipine combination

ARMS (2):
- Telmisartan/Amlodipine, fed (Experimental)
  Interventions: Drug: Telmisartan/Amlodipine; Other: high fat, high caloric meal
- Telmisartan/Amlodipine, fasted (Active Comparator)
  Interventions: Drug: Telmisartan/Amlodipine

INTERVENTIONS:
Drug: Telmisartan/Amlodipine — Fixed dose combination tablet
Other: high fat, high caloric meal
  Arms: Telmisartan/Amlodipine, fed

SUMMARY:
Study to investigate the effect of food intake on the bioavailability of a fixed dose combination of 80 mg telmisartan / 10 mg amlodipine following a high fat breakfast

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥18 and Age ≤55 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial except for oral contraceptives as well as ovary and thyroid hormone replacement
10. Use of drugs which might reasonably influence the results of the trial (especially unspecific inducing agents like St.John´s wort (Hypericum perforatum) or inhibitors like cimetidine) or that prolong the QT/corrected QT interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within one month prior to administration or during the trial
12. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
13. Inability to refrain from smoking during 24 hours prior to dosing and during the trial
14. Alcohol abuse or inability to stop alcoholic beverages for 24 hours prior to dosing and during the trial
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. Any history of relevant low blood pressure
21. Supine blood pressure at screening of systolic <110 mm Hg and diastolic <60 mm Hg
22. History of urticaria
23. History of angioneurotic edema
24. Fructose intolerance

    For female subjects:
25. Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion
26. No adequate contraception during the study and until 1 month of study completion, i.e. implants, injectables, combined oral contraceptives, IUD [intrauterine device], sexual abstinence (for at least 1 month prior to enrolment), vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (incl. hysterectomy). Females, who have not a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide)
27. Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity (AUC0-∞) | up to 168 hours after drug administration
Maximum measured concentration of the analyte in plasma (Cmax) | up to 168 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of telmisartan and amlodipine in plasma over the time interval zero to the last quantifiable data point (AUC0-tz) | up to 168 hours after drug administration
Time from dosing to the maximum concentration in plasma (tmax) | up to 168 hours after drug administration
Terminal rate constant in plasma (λz) | up to 168 hours after drug administration
Terminal half-life in plasma (t1/2) | up to 168 hours after drug administration
Mean residence time in the body after po administration (MRTpo) | up to 168 hours after drug administration
Apparent plasma clearance after p.o. administration (CL/F) | up to 168 hours after drug administration
Apparent volume of distribution during the terminal phase λz after p.o. administration (Vz/F) | up to 168 hours after drug administration
Number of subjects with adverse events | up to 65 days
Assessment of tolerability by investigator on a 4-point scale | day 8 after administration of study drug